CLINICAL TRIAL: NCT05119101
Title: Dexamedtomidine as Adjuvant to Magnesium Sulphate for Intracranial Pressure Control in Pre-eclampsia: a Randomized Controlled Trial.
Brief Title: Dexamedtomidine in Control of Intracranial Pressure in Preeclampsia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Elden Gamal Fakhry, Priniciple investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: intracranial pressure control
Record Dates: First submitted 2021-11-02; First posted 2021-11-12 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Intracranial Pressure Control in Pre-eclampsia
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulphate (Active Comparator): patients will recieve Mg sulphate as loading dose of 4 g diluted in 200 ml normal saline intravenous over 10 minutes followed by 1 g/h infusion for 24 h.
  Interventions: Drug: Magnesium sulfate
- Dexamedotomidine adjuvant to Magnesium sulphate (Active Comparator): Patients will reccieve Mg sulphate as loading dose of 4 g diluted in 200 ml normal saline intravenous over 10 minutes followed by 1 g/h infusion for 24 h. in addition they will receive an intravenous infusion of dexmedetomidine .5 μg/kg diluted in 200 ml normal saline intravenous over 10 minutes followed by .15 μg/kg/hr infusion for 24 h.
  Interventions: Drug: Dexamedotomidine added to Magnesium sulfate

INTERVENTIONS:
Drug: Dexamedotomidine added to Magnesium sulfate — we will give dexamedotomidine and mg sulphate and then measure intracranial pressure at different intervals by measuring Optic nerve sheath diameter (ONSD).
  Other Names: Precedex
  Arms: Dexamedotomidine adjuvant to Magnesium sulphate
Drug: Magnesium sulfate — we will give mg sulphate and then measure intracranial pressure at different intervals by measuring Optic nerve sheath diameter (ONSD).
  Other Names: Mgso4
  Arms: Magnesium sulphate

SUMMARY:
The present study is designed to evaluate the differences in the effect of Mg sulphate alone and dexmedetomidine as an adjuvant to Mg sulphate on intracranial pressure when administered intravenously in cases of pre-eclampsia

DETAILED DESCRIPTION:
Preeclampsia remains one of the leading causes of maternal morbidity and mortality in pregnant women. preeclampsia occurs in 7% to 8% of pregnancies. Preeclampsia is a multisystem progressive disorder characterized by the new onset of hypertension and proteinuria or the new onset of hypertension and significant end-organ dysfunction with or without proteinuria after 20 weeks of gestation or postpartum. Preeclampsia is a potentially severe disease associated with maternal complications. Cerebral oedema is predominantly vasogenic and may be related to failure of cerebral autoregulation with subsequent hyperperfusion, blood brain barrier disruption, and endothelial cell dysfunction.

The optic nerve with its dural sheath cover is considered a window to central nervous system. The subarachnoid space surrounds the optic nerve and communicates freely with the cerebral subarachnoid space. Changes in the optic nerve sheath diameter (ONSD) mirror the changes in the ICP as increases in the ONSD correlates with increase in the ICP.

Magnesium sulphate (MgSO4) is a drug that is routinely used in the treatment of preeclampsia and prevention of eclamptic fits. Currently, several mechanisms have been proposed by researchers to explain the neuroprotective effect of MgSO4 .Dexmedetomidine is a potent alpha-2 adrenergic receptor agonist. dexmedetomidine-induced stimulation of postsynaptic alpha-2 adrenergic receptor on the cerebral blood vessels can cause cerebral vasoconstriction and decrease cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 25-43 and the gestational age above 34 weeks, with diagnostic preeclampsia (Hypertension and proteinuria) occurring after the 20th week of gestation and cesarian section is indicated with systolic blood pressure above 160 and diastolic blood pressure above 100.albumin in urine ++ or +++. No cardiac, hepatic,renal nor neurological problems.

Exclusion Criteria:

1. Age: younger than 25 or older than 43.
2. Pregnant females with mild preeclampsia.
3. Patients with cerebro-vascular diseases, Glaucoma, Hepatic failure, Renal failure .
4. patient who got their MgSO4 medication before the first reading of Optic nerve sheath diameter ONSD were also excluded.
5. History of allergy to dexamedotomidine.

   -

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
will be Optic nerve sheath diameter (ONSD) changes by using ultrasound as an indicator for changes in intracranial pressure in response to treatment with either mg sulphate alone or dexamedotomidine as an adjuvant to mg sulphate. | till two hours after cesarian section

SECONDARY OUTCOMES:
o changes in levels of interleukin 6 (IL-6) in plasma before and after start of treatment in response to any change in brain activity | two hours after cesarian section
o The difference in umbilical blood flow indices by Doppler. | two hours after cesarian section

CONTACTS AND LOCATIONS:
Overall Officials: HossamElden G Fakhry, DR, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes